CLINICAL TRIAL: NCT01000259
Title: Validation of Tumor-Infiltrating T-Cells as a Biomarker for Advanced Epithelial Ovarian Cancer
Brief Title: Study of Tumor Tissue Samples From Patients Who Have Undergone Surgery for Advanced Stage III or Stage IV Ovarian Epithelial Cancer
Status: Recruiting | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-8005; NCI-2011-02279 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-8005; CDR0000391277; GOG-8005 (Other: Gynecologic Oncology Group); GOG-8005 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Stage IIIA Ovarian Cancer; Stage IIIB Ovarian Cancer; Stage IIIC Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

GROUPS / COHORTS (1):
- Ancillary-Correlative: Previously collected tumor tissue samples are analyzed for TIL via immunohistochemistry and double immunofluorescence assays using standard immunostaining.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Samples are analyzed in laboratory studies

SUMMARY:
This research study is looking at tumor tissue samples from patients who have undergone surgery for advanced stage III or stage IV ovarian epithelial cancer. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn how tumor infiltrating T cells can predict how patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To validate the ability of intratumoral tumor-infiltrating T lymphocytes (TILs) to predict progression-free survival (PFS) in patients with suboptimally debulked advanced stage III or IV ovarian epithelial cancer.

II. To validate the ability of intratumoral TILs to predict PFS in patients with optimally debulked disease.

SECONDARY OBJECTIVES:

I. To validate the ability of intratumoral TILs to predict overall survival of patients with suboptimally debulked disease.

II. To validate the ability of intratumoral TILs to predict overall survival of patients with optimally debulked disease.

OUTLINE:

Patients are stratified according to status of debulked disease (suboptimal vs optimal).

Previously collected tumor tissue samples are analyzed for tumor-infiltrating lymphocytes (TIL) via immunohistochemistry and double immunofluorescence assays using standard immunostaining.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III or IV ovarian epithelial cancer and enrolled on Gynecologic Oncology Group (GOG)-0136 and a GOG front-line platinum/taxol chemotherapy trial (GOG-0114, GOG-132, GOG-0158, or GOG-0162)
* Must have fixed and paraffin-embedded tissue from primary surgery available from 1 of the following sources:

  * Patients enrolled on GOG-0136 and a GOG front-line platinum/taxol chemotherapy trial(GOG-0114, GOG-0132, GOG-0158, and GOG-0162)
  * Patients who have had either optimal or suboptimal cytoreductive surgery
  * Patients for whom adequate demographic data, including major prognostic factors and follow-up information, were collected
* Evaluable patients must have had measurable or nonmeasurable disease
* Demographic and follow-up data available

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2004-09; Primary Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival curves | Baseline
  The Kaplan-Meier method will be used to estimate the survival curves, and the log-rank test will be used to test the difference between survival curves for TIL positive and negative patients. All of the tests will be two-sided and the significant levels will be set a 0.05.
Progression-free survival curves | Baseline
  The Kaplan-Meier method will be used to estimate the survival curves, and the log-rank test will be used to test the difference between survival curves for TIL positive and negative patients. All of the tests will be two-sided and the significant levels will be set a 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: George Coukos, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States